CLINICAL TRIAL: NCT03114501
Title: Dyadic Yoga Intervention for Patient With Head and Neck Cancer Undergoing Radiotherapy and Their Family Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1127; NCI-2018-01163 (Other: NCI CTRP)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasms of Lip Oral Cavity and Pharynx; Head and Neck Cancer
Keywords: Malignant neoplasms of lip oral cavity and pharynx; Head and Neck Cancer; Yoga; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Yoga; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Program Group (Experimental): Participants take part in the partner-based yoga program.
  Questionnaire completed during each week of radiation therapy about participant's feelings about the yoga sessions.
  Questionnaires completed before first radiation treatment, during week 3 of radiation therapy, and again after completion of treatment schedule (usually 6 weeks later).
  Interventions: Behavioral: Yoga; Behavioral: Yoga Questionnaire; Behavioral: Symptom Questionnaires
- Waitlist Control Group (WLC) (Experimental): Participants receive standard of care.
  Questionnaires completed before first radiation treatment, during week 3 of radiation therapy, and again after completion of treatment schedule (usually 6 weeks later).
  After the study has been completed, participant and caregiver/alternative caregiver offered the opportunity to take part in the partner-based yoga program.
  Interventions: Behavioral: Symptom Questionnaires

INTERVENTIONS:
Behavioral: Yoga — Participants receive yoga sessions up to 5 days per week, based on the patient's schedule, over the course of patients' Radiation Therapy (up to 15 sessions, 45-60 min. each). Yoga sessions audio and video recorded.
  Arms: Yoga Program Group
Behavioral: Yoga Questionnaire — Questionnaire completed during each week of radiation therapy about participant's feelings about the yoga sessions.
  Other Names: Survey
  Arms: Yoga Program Group
Behavioral: Symptom Questionnaires — Symptom questionnaires completed before first radiation treatment, during week 3 of radiation therapy, and again after completion of treatment schedule (usually 6 weeks later).
  Other Names: Surveys

SUMMARY:
Objectives:

Primary Aim:

Examine the feasibility of a dyadic yoga program in 40 Head and Neck Cancer (HNC) patients undergoing radiotherapy (RT) and their family caregivers.

Secondary Aims:

1. Establish the initial efficacy of the yoga program in patients and their caregivers regarding quality of life (QOL) outcomes (i.e., fatigue, sleep disturbance, depressive symptoms, and overall QOL) and objective performance outcomes (i.e, sit to stand test and grip strength).

DETAILED DESCRIPTION:
Caregiver:

If you agree to take part in this study, your demographic information (such as your age, sex, and race) will be recorded at your first visit.

After your first visit, you and the patient will be assigned to 1 of 2 groups. You will either automatically be assigned to Group 1 if you are in the first 10 couples to join the study, or you will be randomly assigned (as in the roll of dice) to Group 1 or Group 2.

This random assignment is done because no one knows if one study group is better, the same, or worse than the other group. You have about an equal chance of being assigned to each group. However, the assignment is also based on other factors such as age and disease status.

If you are in Group 1, you will take part in the partner-based yoga program.

If you are in Group 2, you will not take part in the partner-based yoga program but will complete the same questionnaires as Group 1. After the study has been completed, you and the patient will be offered the opportunity to take part in the partner-based yoga program. This will be offered outside the study and will be offered at no cost to you.

Group 1 - Yoga Sessions and Alternate Caregiver Questionnaire:

If you are in Group 1, you will take part in up to 15 sessions of yoga over the course of the patient's radiation therapy. Each 45- to 60-minute session will be guided by an instructor either face-to-face or by videoconferencing (FaceTime). You should attend each session together as partners.

If you do not have access to a personal handheld device (such as an iPhone or iPad), an iPad will be assigned to you. You will be asked to complete an iPad agreement form and return the iPad on the date that is noted in the agreement. If the device breaks, please tell the study staff right away.

During the yoga sessions, you will be asked to do deep-breathing exercises and perform different stretching and movement exercises. The movements are designed not to be difficult, and you will sit on the floor or in a chair while you do them. You can move through the exercises at your own pace. The instructor will be available to answer any questions you may have about the practice of yoga.

The yoga sessions may be audio- and video-recorded. This is so the researchers can keep track of the quality of the sessions. Only the study staff will be able to review this tape. The audio and video files are digital and will be destroyed after 7 years. If you do not allow the sessions to be audio- or video-recorded, you cannot take part in this study.

At your fifth session, you will be given a DVD and instructions for practicing yoga at home. While the patient is receiving radiation therapy, you will be asked to practice at home 1 time a day either with the patient or alone on the days you do not have a session at the clinic.

During each week of radiation therapy, you will also complete a questionnaire on your feelings about the yoga sessions. You will be asked to list what you liked or disliked, what you found most and least useful, and how you would rate the instructor. You will also be asked about how often you practice yoga outside of class and if you think you are benefitting from the yoga program. It should take about 5 minutes to answer this questionnaire. Your answers to the questions will not be shared with the patient.

If you are an alternate caregiver, you will complete a quality-of-life questionnaire at your first yoga session and at the end of the patient's treatment. The questionnaire at the end of treatment can be completed by mail, over the phone with the study staff, or at a clinic session. Completing the questionnaire should take less than 10 minutes.

Groups 1 and 2 - Questionnaires:

You will complete about 12 questionnaires before the patient's first radiation treatment) and again 3 months later. The questionnaires ask about your health, any symptoms you may be having, your mood, fatigue level, sleeping habits, relationship, health care, work productivity, and quality of life. It should take about 55 minutes to complete these questionnaires.

During the last week of the patient's radiation therapy, you will complete about 8 questionnaires. The questionnaires ask about your health, any symptoms you may be having, your mood, fatigue level, sleeping habits, relationship, and quality of life. It should take about 45 minutes to complete these questionnaires.

Length of Study:

Your participation on this study will be over when you have completed the last questionnaires.

Patient:

If you agree to take part in this study, your medical history and demographic information (such as your age, sex, and race) will be recorded at your first visit. Additional medical information will be collected from your medical record, such as current/past nicotine use.

If you sign this consent, your caregiver will be approached to take part in this study.

After your first visit, you and your caregiver will be assigned to 1 of 2 groups. You will either automatically be assigned to Group 1 if you are in the first 10 couples to join the study, or you will be randomly assigned (as in the roll of dice) to Group 1 or Group 2.

This random assignment is done because no one knows if one study group is better, the same, or worse than the other group. You have about an equal chance of being assigned to each group. However, the assignment is also based on other factors such as your age and the status of the disease.

If you are in Group 1, you will take part in the partner-based yoga program.

If you are in Group 2, you will not take part in the partner-based yoga program but will complete the same questionnaires as Group 1. After the study has been completed, you and your caregiver/alternative caregiver will be offered the opportunity to take part in the partner-based yoga program.

Group 1 - Yoga Sessions:

If you are in Group 1, you will take part in up to 15 sessions of yoga over the course of radiation therapy. Each 45- to 60-minute session will be guided by an instructor either face-to-face or by videoconferencing (FaceTime). You should attend each session together as partners.

If you do not have access to a personal handheld device (such as an iPhone or iPad), an iPad will be assigned to you. You will be asked to complete an iPad agreement form and return the iPad on the date that is noted in the agreement. If the device breaks, please tell the study staff right away.

During the yoga sessions, you will be asked to do deep-breathing exercises and perform different stretching and movement exercises. The movements are designed not to be difficult, and you will sit on the floor or in a chair while you do them. You can move through the exercises at your own pace. The instructor will be available to answer any questions you may have about the practice of yoga.

The yoga sessions may be audio- and video recorded. This is so the researchers can keep track of the quality of the sessions. Only the study staff will be able to review this tape. The audio and video files are digital and will be destroyed after 7 years. If you do not allow the sessions to be audio- or video-recorded, you cannot take part in this study.

At your fifth session, you will be given a DVD and instructions for practicing yoga at home. While you are receiving radiation therapy, you will be asked to practice at home 1 time a day either with your caregiver or alone on the days you do not have a session at the clinic.

During each week of radiation therapy, you will also complete a questionnaire on your feelings about the yoga sessions. You will be asked to list what you liked or disliked, what you found most and least useful, and how you would rate the instructor. You will also be asked about how often you practice yoga outside of class and if you think you are benefitting from the yoga program. It should take about 5 minutes to answer this questionnaire. Your answers to the questions will not be shared with your caregiver.

Groups 1 and 2 - Questionnaires:

You will complete about 12 questionnaires before your first radiation treatment and again 3 months later The questionnaires ask about your health, any symptoms you may be having, your mood, fatigue level, sleeping habits, relationship, health care, work productivity, and quality of life. It should take about 55 minutes to complete these questionnaires.

During your last week of radiation therapy, you will complete about 8 questionnaires. The questionnaires ask about your health, any symptoms you may be having, your mood, fatigue level, sleeping habits, relationship, and quality of life. It should take about 45 minutes to complete these questionnaires.

During Week 3 of radiation therapy and 4 weeks after radiation therapy, you will complete the symptom questionnaire. It should take about 5 minutes to complete. You can complete it over the phone with the study staff or at a clinic session.

Additional Tests for Both Groups:

You will complete a sit-to-stand and grip strength test before your first radiation treatment and once weekly at radiation therapy visits during the time that you receive radiation therapy. The sit-to-stand test measures how easily you sit down and stand up out of a chair. The grip strength test measures the strength of your hands and lower arms. These tests should take about 5 minutes to complete.

Length of Study:

Your participation on this study will be over when you have completed the last questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. (Patients) Diagnosed with a primary HNC and going to receive at least 4 weeks of RT with at least 20 fractions
2. (Patients) ECOG performance status of 2 or lower
3. (Patients) having an informal family caregiver (spouse, romantic partner, adult child, or sibling) who is willing to participate. If patients do not have one consistent primary caregiver for the duration of the study, they may be accompanied to the yoga sessions by an alternate caregiver who meets eligibility criteria.
4. (Patients) having a smart phone (phase 2 only)
5. (Patients and Caregivers) must be (1) at least 18 years old
6. (Patients and Caregivers) able to read and speak English
7. (Patients and Caregivers) able to provide informed consent

Exclusion Criteria:

1. (Patients) regularly (self-defined) participated in a yoga practice in the year prior to diagnosis
2. (Patients) cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team
3. (Patients and Caregivers) those who participate in phase 1 are ineligible to participate in phase 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a Dyadic Yoga Program in Head and Neck Cancer (HNC) Participants Undergoing Radiotherapy (RT) | 6 weeks after radiation therapy
  Trial considered feasible if 1) ≥ 50% of eligible couples consent (i.e., approach 80 couples to obtain 40 consents); 2) ≥ 70% of enrolled couples complete both assessments; 3) on average ≥ 50% of all practice sessions are attended.

SECONDARY OUTCOMES:
Efficacy of a Dyadic Yoga Program in Head and Neck Cancer (HNC) Participants Undergoing Radiotherapy (RT) | 6 weeks after radiation therapy
  Efficacy of the yoga program determined by responses on quality of life (QOL) questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, MA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org